CLINICAL TRIAL: NCT06209918
Title: Effect of Bioptron Light Therapy on Pregnancy Related Carpal Tunnel Syndrome
Brief Title: Effect of Bioptron Light on Carpal Tunnel Syndrome(BLCTS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Magdy Ahmed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003875
Record Dates: First submitted 2023-07-21; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Carpal Tunnel Syndrome Pregnancy
Keywords: Bioptron light therapy; Phototherapy; Carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group that recieve bioptron light and advice and patient education (Experimental): patients will recieve bioptron light therapy for 10 minutes per session, 3 sessions per week, for 4 weeks.
  Interventions: Device: bioptron light therapy
- control group that recieve advice and patient education and wrist brace (Other): will keep the wrist in a neutral position, not bent back or bent down too far
  Interventions: Device: wrist brace

INTERVENTIONS:
Device: bioptron light therapy — patient will be sitting on comfortable chair with the hand placed on an armrest in an extended and supinated position. Firstly, the skin over the wrist area will be exposed and cleaned by alcohol to achieve maximal penetration of light. Then, the bioptron device will be held perpendicular to the surface of the treated area, at a distance of 10 cm.
  Arms: group that recieve bioptron light and advice and patient education
Device: wrist brace — will keep the wrist in a neutral position, not bent back or bent down too far
  Arms: control group that recieve advice and patient education and wrist brace

SUMMARY:
The purpose of this study is to investigate the effect of bioptron light therapy on pregnancy related carpal tunnel syndrome

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is a symptomatic compression neuropathy of the median nerve at the level of the wrist, characterized by hand pain, numbness, and tingling in the distribution of the median nerve (thumb, index, middle finger, and the radial side of the ring finger) and a reduction in grip strength and hand function. The severity of symptoms can be clinically categorized into mild, moderate, and severe Bioptron phototherapy acts as a "sterile" trigger on human in vitro isolated peripheral blood mononuclear cells (PBMCs), affecting their cytokine production and driving the immune response towards an anti-inflammatory/reparative profile and representing a non-pharmaceutical and non-invasive option for several clinical conditionsA randomized control study, the women will be randomly assigned into two groups, (31 women for each group) equal in number. Group (A) will include 31 women will receive Bioptron light combined with advice and patient education (10 minutes per session, 3 sessions per week, for 4 weeks). Group (B) will be receiving advice only for same duration as group (A)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females clinically daignosed with carpal tunnel syndrome at least 1 month
* age will range from (25-35) years.
* body mass index (BMI) will be (BMI ≤ 35 kg/m2)

Exclusion Criteria:

* history of neurologic disease
* hand surgery
* hand trauma,
* diabetes mellitus
* cervical spondylosis
* osteoarthritis of cervical spine and wrist joint
* chronic renal failure
* heart failure
* connective tissue disorders

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women having carpal tunnel syndrome
Enrollment: 62 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Nerve conduction studies (NCS) | 4 weeks
  assess sensory and motor nerve conduction velocity,gf and sensory nerve action potential

SECONDARY OUTCOMES:
Visual analogue scale | 4 weeks
  assess pain intensity

OTHER OUTCOMES:
Boston carpal tunnel questionnaire | 4 weeks
  Assess Symptom severity and functional capacity

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ma Ahmed, lecturer, Principal Investigator — Cairo University
Locations (1):
- Sara Magdy Ahmed, Giza, Egypt